CLINICAL TRIAL: NCT00843557
Title: Impact of Gender on Hospitalized Patients
Status: Completed | Type: Observational
Sponsor: University of Virginia (Other)
Collaborators: Vanderbilt University (Other)
Responsible Party: Robert G. Sawyer MD, Universtiy of Virginia
Other Study IDs: 9481; 00170560
Record Dates: First submitted 2009-02-12; First posted 2009-02-13 (Estimated); Last update posted 2016-10-27 (Estimated); Status verified 2016-10

CONDITIONS: Critical Illness
Keywords: critical illness; intensive care; nosocomial infection
MeSH Terms: conditions — Critical Illness; Cross Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- all ICU admissions: patients admitted to the ICU for greater then 72hrs

SUMMARY:
The purpose of this study is to better understand the relationship between gender (being a man or a woman), infections caught in the hospital, and serious illness. Five hundred seventy patients 18 years of age or older who are critically (seriously) ill and admitted to the Intensive Care Unit (ICU) for at least 48 hours will participate in this study. Patients will be studied while receiving regular ICU treatment according to local standards. Blood specimens will come from patients either as wasted blood (University of Virginia) or blood collected from patients specifically for the study (Vanderbilt University). All patients will be followed daily until death or discharge from the ICU. The researchers believe that they will find a similar risk of infection for men and women overall.

DETAILED DESCRIPTION:
The purpose of this study is to gain knowledge that will be used to design further interventional studies to better define beneficial therapies related to gender, infection, and critical illness, such as modulation of hormone levels in a sex-specific manner. This is a two-year observational study in which approximately a total of 570 patients will be enrolled. All patients will be 18 years of age or older and admitted to the Intensive Care Unit (ICU) for at least 48 hours. Patients will be studied while receiving accepted and approved therapy according to local standards. Data obtained will be that which would normally be considered part of a standard complete medical history. Specimens will come from patients either as wasted blood (University of Virginia) or blood drawn from patients specifically for this purpose (Vanderbilt University). The maximum blood removed will be 30 ml twice weekly and is considered a minor risk. All specimens analyzed, regardless of institution, are done so in a blinded manner, identified only by study number and specimen number or through password and encryption protected servers when communicated electronically. Since the cohort is comprised of all patients admitted to an ICU, recruitment in the normal sense is not practical. An initial comparison of demographic data, severity of illness, frequency of comorbidities, hormone and cytokine levels, and outcome variables will be compared between males and females treated for infection. All patients will be followed daily until death or discharge from the ICU. It is anticipated that a similar risk of infection for men and women overall will be determined. Specific Aim I of the study is to prospectively determine and compare the incidence of and associated mortality from hospital-acquired infections in a large, critically-ill population of pre-menopausal women, post-menopausal women, and men after controlling for multiple pre-defined confounding variables. The Specific Aim II of the study is to determine the relationship between sex hormonal status, systemic cytokine levels, and the incidence of and outcome from hospital-acquired infections, as well as the relative contribution of infection and end-of-life decisions to outcome in subjects dying under study.

ELIGIBILITY:
Inclusion Criteria:Inclusion Criteria:

1. All patients >= 18 years old admitted to the ICU for >= 48 hours.

Exclusion Criteria:

1. Age < 18 years old.
2. Death or discharge within 48 hours of ICU admission.
3. Patients not on a surgical service.
4. Patients admitted with a primary diagnosis of burns.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to general surgery and trauma ICU
Sampling Method: Non-Probability Sample
Enrollment: 2400 (Actual)
Dates: Start 2001-09; Primary Completion 2006-05 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Death following admission to the ICU | duration of hospitalization

SECONDARY OUTCOMES:
incidence of infection of patients treated in the ICU | duration of hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Robert G Sawyer, MD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States